CLINICAL TRIAL: NCT00997945
Title: A Phase I, Open-label, Single-arm Study to Determine the Single and Multiple Dose Pharmacokinetics of 10mg ZD4054 (Zibotentan) Administered Once Daily in Male, Elderly Chinese Patients With Advanced Solid Malignancies
Brief Title: 10mg ZD4054 (Zibotentan) PK Study in Male, Elderly Chinese Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D4320C00041
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Advanced Solid Malignancies
Keywords: Phase I, advanced solid malignancies, advance solid tumour; advanced cancer; ZD4054 (Zibotentan); china; PK; pharmacokinetics
MeSH Terms: interventions — ZD4054

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): ZD4054 (Zibotentan) 10mg
  Interventions: Drug: ZD4054 (Zibotentan)

INTERVENTIONS:
Drug: ZD4054 (Zibotentan) — 10 mg ZD4054 (Zibotentan) once daily on Day1, Day4 to Day15
  Other Names: Zibotentan

SUMMARY:
The purpose of this study is to assess the pharmacokinetics of single and multiple doses of 10mg ZD4054 (Zibotentan) in male, elderly Chinese patients with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Histological and/or cytological confirmed advanced solid malignancies
* WHO performance status<2

Exclusion Criteria:

* History of significant gastrointestinal impairment, as judged by the investigator, that could significantly affect the absorption of ZD4054 (Zibotentan) , including the ability to swallow the tablet whole.
* ALT or AST³2.5 ´ULRR. If liver metastases are present ALT or AST more than 5times ULRR, Serum bilirubin > 1.5 x ULRR, Serum creatinine>1.5 x ULRR or creatinine clearance of <50mL/min calculated by Cockroft-Gault
* Recent (<14 days) major surgery prior to entry into the study, or a surgical incision that is not fully healed, Radical radiotherapy within the previous 4 weeks, or unresolved acute or subacute toxicities from prior radiotherapy

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetics of single and multiple doses of 10mg ZD4054 (Zibotentan) in male, elderly Chinese patients with advanced solid malignancies | PK samples will be taken until Day 16

SECONDARY OUTCOMES:
To assess the safety and tolerability of single and multiple doses of 10mg ZD4054 (Zibotentan) in male, elderly Chinese patients with advanced solid malignancies | Safety assessments to be taken until Day 16 (while patient remains on study treatment), then every 8 weeks until treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Li Jin, Principal Investigator — The Cancer Hospital Affiliated Fudan University; Helen Lin, Study Director — AstraZeneca China MC
Locations (1):
- Research Site, Shanghai, Shanghai Municipality, China